CLINICAL TRIAL: NCT06379347
Title: HOspitalized Patients and Clinical flUid Status, Assessment Using Point Of Care UltraSound
Acronym: HOCUS-POCUS
Status: Recruiting | Type: Observational
Sponsor: Flevoziekenhuis (Other)
Responsible Party: Sponsor
Other Study IDs: FZ 23/41
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Volume Status

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: POCUS performed on clinical indication — POCUS performed on clinical indication

SUMMARY:
Point of care ultrasound (POCUS) of the inferior vena cava (IVC) is a tool for assessing volume status through ultrasonography. Using a point of care ultrasound device, the physician can perform an ultrasound of the vena cava at the bedside. Previous research has demonstrated a correlation between right atrial pressure and the vena cava's diameter. Nonetheless, the majority of research has been conducted in critically ill populations to predict fluid responsiveness in patients with more complex hemodynamics. There is limited data available on the value of IVC ultrasound in the sub-acute setting on the regular ward for clinical decision-making regarding whether a patient is hypovolemic or hypervolemic. This study's objective is to assess the diagnostic utility of point-of-care ultrasonography of the IVC, by using a standardized methodology, performed by qualified ward physicians in a conventional nursing ward.

DETAILED DESCRIPTION:
The study will be carried out on patients over the age of 18 who were admitted to the general ward between for at least 24 hours and who had a clinical indication for an IVC ultrasound. Patients are informed through an informed consent form and are given the opportunity to opt-out. When there are no objections, the patient's data is collected for the study. Patients who are using vasopressors at the time of the ultrasound are excluded from the study. In addition, patients who require invasive or non-invasive ventilation (optiflow, CPAP, BPAP) are also excluded.

The ultrasounds are performed by trained physicians based on a standard operating procedure. The longitudinal portion of the IVC is scanned and a cine loop of 10 seconds is made during a respiratory cycle to determine the diameter of the IVC (dIVC). After the recording is paused, the dIVC will be measured 2 cm caudal to the junction of the hepatic vein and IVC to standardize the measurements. Measurements are taken at peak expiration (dIVCe) and inspiration (dIVCi) by measuring the vein lumen at one respiratory cycle from one interior wall to the opposite interior wall.

Data is collected at the time of admission and after 48 hours (or prematurely if the patient is discharged). During the initial assessment, the patient's demographics, clinical data, physical examination, vitals , laboratory parameters, and the POCUS IVC (minimal and maximal diameter, percentage collapse) are registered. The Charlson Comorbidity Index is used to quantify the severity of comorbidities in the patients. Additionally, the patient's overall health status is measured by the ECOG Performance Status Scale.

Once the initial measurements are done, a clinical diagnosis of the patient's volume status will be established. 48 hours later, more data will be gathered for the follow-up. The data includes vitals and laboratory parameters. It is also noted whether the POCUS influenced the management of treatment (IV fluid or diuretic therapy) of each patient. Following this assessment, a clinical diagnosis in retrospect at the time of the ultrasound at baseline about the volume status is established.

The diagnostic accuracy for hypovolemia and hypervolemia cases are analyzed. The sensitivity, specificity, positive predictive value, and negative predictive value are also determined. Furthermore, the area under the curve (AUC) for hypo- and hypervolemia were computed.

A descriptive analysis of the changes over time will be carried out in the subgroup with follow-up measurements. The interpretation of the images at the time of the ultrasound serves as the foundation for the main analysis. A second assessor will verify the images retrospectively in a subset, recalculating the diameter and evaluating their quality. A descriptive analysis will be conducted on the quality of measurements. Moreover, an exploratory analysis will be carried out to ascertain the best location and cutoff points for identifying volume status.

ELIGIBILITY:
Inclusion Criteria:

* Patient is over 18 years old.
* Patient has a clinical indication for making a IVC ultrasound.
* Patient is admitted until at least 24 hours after the first ultrasound.

Exclusion Criteria:

* Patients who are using vasopressors at the time of the ultrasound.
* Patients who require invasive or non-invasive (optiflow, CPAP, BPAP) ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the general ward with a clinical indication for performing VCI ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Volume status | 48 hours
  Depleted, overloaded, or normal volume status at baseline, determined 48 hours after performing the ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Koen de Heer, MD PhD, Principal Investigator — Flevoziekenhuis
Locations (1):
- Flevoziekenhuis, Almere Stad, Netherlands

REFERENCES:
- [Background] Kircher BJ, Himelman RB, Schiller NB. Noninvasive estimation of right atrial pressure from the inspiratory collapse of the inferior vena cava. Am J Cardiol. 1990 Aug 15;66(4):493-6. doi: 10.1016/0002-9149(90)90711-9. PMID 2386120